CLINICAL TRIAL: NCT03047941
Title: Determination of Optimal Cutoff Value of 4 Tests (DES-OSA, STOP-Bang, OSA50, P-SAP) for Screening Severe Hypoxemic OSA (Obstructive Sleep Apnea) Patients
Brief Title: Determination of Optimal Cutoff Value for Screening Severe Hypoxemic OSA (Obstructive Sleep Apnea) Patients
Status: Withdrawn | Type: Observational
Why Stopped: Lack of participants
Sponsor: Astes (Other)
Responsible Party: Principal Investigator, Eric DEFLANDRE, MD, PhD, FCCP, FAHA, Principal Investigators, Astes
Other Study IDs: REES2
Record Dates: First submitted 2017-02-06; First posted 2017-02-09 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All patients: All patients included in the present study
  Interventions: Diagnostic Test: Determination of optimal cutoff values.

INTERVENTIONS:
Diagnostic Test: Determination of optimal cutoff values. — The results of the four scores will be compared with the results of the polysomnography (PSG). A statistical analysis will be performed to determine the optimal cutoff value of each of the four scores to detect severe OSA patient with hypoxemia.

SUMMARY:
The 4 following scores have been proposed to detect OSA (Obstructive Sleep Apnea): DES-OSA, STOP-Bang, P-SAP, and OSA50.

The aim of this study is to evaluate the optimal cutoff value of these four scores to detect specifically serve OSA patients with hypoxemia.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled to have a PSG in the sleep laboratory center.

Exclusion Criteria:

* Patients < 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients scheduled to have a PSG in the sleep laboratory center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
Adequacy of STOP-Bang to detect severe hypoxemic OSA patients | One week.
  Adequacy of STOP-Bang after comparison with the results of the PSG.
Adequacy of P-SAP to detect severe hypoxemic OSA patients | One week
  Adequacy of P-SAP after comparison with the results of the PSG.
Adequacy of OSA50 to detect severe hypoxemic OSA patients | One week
  Adequacy of OSA50 after comparison with the results of the PSG.
Adequacy of DES-OSA to detect severe hypoxemic OSA patients | One week
  Adequacy of DES-OSA after comparison with the results of the PSG.

CONTACTS AND LOCATIONS:
Locations (1):
- ASTES, Bouge, Namur, Belgium

IPD SHARING:
Plan to Share IPD: No